

# GİRİŞİMSEL OLMAYAN KLİNİK ARAŞTIRMALAR ETİK KURULU

# ERİŞKİN HASTALAR İÇİN BİLGİLENDİRİLMİŞ GÖNÜLLÜ OLUR FORMU

Araştırma Projesinin Adı: Yağ Çekme Terapisinin Diş Ve Dişeti Sağlığı Üzerine Etkisinin

Değerlendirilmesi

Sorumlu Araştırıcının Adı: Dr. Öğr. Ü. Tuğba AYDIN

Diğer Araştırıcıların Adı: Arş. Gör. Ahmet Bedreddin ŞAHİN

Destekleyici (varsa):

"Yağ Çekme Terapisinin Diş Ve Dişeti Sağlığı Üzerine Etkisinin Değerlendirilmesi" isimli bir çalışmada yer almak üzere davet edilmiş bulunmaktasınız. Bu çalışma, araştırma amaçlı olarak yapılmaktadır ve katılım gönüllülük esasına dayalıdır. Çalışmaya katılma konusunda karar vermeden önce araştırma hakkında sizi bilgilendirmek istiyoruz. Çalışma hakkında tam olarak bilgi sahibi olduktan sonra ve sorularınız cevaplandıktan sonra eğer katılmak isterseniz sizden bu formu imzalamanız istenecektir. Bu araştırma, Atatürk Üniversitesi Diş Hekimliği Fakültesi Periodontoloji Anabilim Dalı'nda, Dr. Tuğba AYDIN sorumluluğu altındadır.

# Çalışmanın amacı nedir; benden başka kaç kişi bu çalışmaya katılacak?

Çalışmaya toplam 100 birey alınması planlanmaktadır. Bu çalışmada, klorheksidin glukonat içeren gargaraların ve çeşitli yağlarla yapılan yağ çekme terapisinin birbiriyle ve kendi aralarında, dişteki ve dişetindeki etkilerinin karşılaştırılması ve birbirlerine karşı üstünlüklerinin belirlenmesi amaçlanmaktadır

### Bu çalışmaya katılmalı mıyım? (Bu bölüm aynen korunacaktır)

Bu çalışmada yer alıp almamak tamamen size bağlıdır. Şu anda bu formu imzalasanız bile istediğiniz herhangi bir zamanda bir neden göstermeksizin çalışmayı bırakmakta özgürsünüz. Eğer katılmak istemez iseniz veya çalışmadan ayrılırsanız, doktorunuz tarafından sizin için en uygun tedavi planı uygulanacaktır. Aynı şekilde çalışmayı yürüten doktor çalışmaya devam etmenizin sizin için yararlı olmayacağına karar verebilir ve sizi çalışma dışı bırakabilir, bu durumda da sizin için en uygun tedavi seçilecektir.

### Bu çalışmaya katılırsam beni ne bekliyor?

Öncelikle diş taşı temizliği ve polisaj yapılacak, oral hijyen eğitimi verilecektir. İki haftalık hazırlık periyodunda mekanik plak temizliğinin tam yapılması gerekmektedir.

İki haftalık hazırlık periyodu sonrası kontrol muayenesi yapılacak ve dijital spektrofotometre ile diş rengi tayini yapılacaktır.

Daha sonra katılımcılara, klorheksidin içeren ağız gargarası veya çörek otu yağı, hindistan cevizi yağı ve menengiç yağı arasından biri 4 gün boyunca mekanik plak temizliği yapılmadan kullandırılacaktır. 4 günün sonunda diş eti oluğu kanama indeksi, Quigley-Hein ve Turesky plak indeksi ve dijital spektrofotometre ile diş rengine tekrar bakılacak ve kullanılan ürünle ilgili memnuniyet ölçecek anket yapılacaktır. Sonuçlar değerlendirilecektir.

#### Calışmanın riskleri ve rahatsızlıkları var mıdır?

Yapılan uygulamalarda fiziksel sağlığınıza zarar verecek herhangi bir risk unsuru bulunmamaktadır.

| BGOF-Girişimsel olmayan-Erişkin | Rev. Tarihi / No.su: | Sayfa |
|---------------------------------|----------------------|-------|
| | 21.11.2019/01 | 1/3 |

# GİRİŞİMSEL OLMAYAN KLİNİK ARAŞTIRMALAR ETİK KURULU

# Çalışmada yer almamın yararları nelerdir?

Çalışmanın tamamlanması durumunda; yağ terapisinin plak temizliğinde etkinliği gösterilirse, plak temizliğinde daha uygun fiyatlı, ulaşılması kolay ve doğal ürünlerin kullanılması sağlanabilir.

### Bu çalışmaya katılmamın maliyeti nedir? (Bu bölüm aynen korunacaktır)

Çalışmaya katılmakla parasal yük altına girmeyeceksiniz ve size de herhangi bir ödeme yapılmayacaktır.

#### Kişisel bilgilerim nasıl kullanılacak? (Bu bölüm aynen korunacaktır)

Çalışma doktorunuz kişisel bilgilerinizi, araştırmayı ve istatiksel analizleri yürütmek için kullanacaktır ancak kimlik bilgileriniz gizli tutulacaktır. Yalnızca gereği halinde, sizinle ilgili bilgileri etik kurullar ya da resmi makamlar inceleyebilir. Çalışmanın sonunda, kendi sonuçlarınızla ilgili bilgi istemeye hakkınız vardır. Çalışma sonuçları çalışma bitiminde tıbbi literatürde yayınlanabilecektir ancak kimliğiniz açıklanmayacaktır.

#### Daha fazla bilgi için kime başvurabilirim?

Çalışma ile ilgili ek bilgiye gereksiniminiz olduğunuzda aşağıdaki kişi ile lütfen iletişime geçiniz.

ADI : Tuğba Aydın GÖREVİ : Dr. Öğr. Ü. TELEFON : 442-231 2173

## (Katılımcının/Hastanın Beyanı)

Araştırmaya katılmam konusunda zorlayıcı bir davranışla karşılaşmış değilim. Eğer katılmayı reddedersem, bu durumun tıbbi bakımıma ve hekim ile olan ilişkime herhangi bir zarar getirmeyeceğini de biliyorum. Projenin yürütülmesi sırasında herhangi bir neden göstermeden araştırmadan çekilebilirim. (Ancak araştırmacıları zor durumda bırakmamak için araştırmadan çekileceğimi önceden bildirmemim uygun olacağının bilincindeyim). Ayrıca tıbbi durumuma herhangi bir zarar verilmemesi koşuluyla araştırmacı tarafından araştırma dışı da tutulabilirim.

Araştırma için yapılacak harcamalarla ilgili herhangi bir parasal sorumluluk altına girmiyorum. Bana da bir ödeme yapılmayacaktır.

Araştırmadan elde edilen benimle ilgili kişisel bilgilerin gizliliğinin korunacağını biliyorum.

Araştırma uygulamasından kaynaklanan nedenlerle meydana gelebilecek herhangi bir sağlık sorunumun ortaya çıkması halinde, her türlü tıbbi müdahalenin sağlanacağı konusunda gerekli güvence verildi. (Bu tıbbi müdahalelerle ilgili olarak da parasal bir yük altına girmeyeceğim).

| BGOF-Girişimsel olmayan-Erişkin | DCOF Civisius al alumanas Frielia | Rev. Tarihi / No.su: | Sayfa |
|---|---|---|---|
| | 21.11.2019/01 | 2/3 | |

# GİRİŞİMSEL OLMAYAN KLİNİK ARAŞTIRMALAR ETİK KURULU

Araştırma sırasında bir sağlık sorunu ile karşılaştığımda; herhangi bir saatte, Dr.....(Doktor ismi), .....(telefon ve adres) 'ten arayabileceğimi biliyorum. (Doktor ismi, telefon ve adres bilgileri mutlaka belirtilmelidir)

Bana yapılan tüm açıklamaları ayrıntılarıyla anlamış bulunmaktayım. Bu koşullarla söz konusu klinik araştırmaya kendi rızamla, hiç bir baskı ve zorlama olmaksızın, gönüllülük içerisinde katılmayı kabul ediyorum.

İmzalı bu form kağıdının bir kopyası bana verilecektir.

| Katılımcı |
|----------------|
| Adı, soyadı: |
| Adres: |
| Tel: |
| İmza: |
| Tarih: |
| Görüşme tanığı |
| Adı, soyadı: |
| Adres: |
| Tel: |

Katılımcı ile görüşen hekim

Adı soyadı, unvanı:

Adres:

İmza: Tarih:

Tel: İmza:

Tarih:

AYDINLATMA ve KATILIMCININ BEYANI KESİNLİKLE BİRBİRLERİNİN DEVAMI ŞEKLİNDE OLACAKTIR. AYRI AYRI SAYFALARDA YER <u>ALMAYACAKTIR.</u>

| BGOF-Girişimsel olmayan-Erişkin | Rev. Tarihi / No.su: | Sayfa |
|---------------------------------|----------------------|-------|
| | 21.11.2019/01 | 3/3 |